CLINICAL TRIAL: NCT02651259
Title: A Phase I/II Trial of the Pharmacokinetics, Tolerability, and Safety of Once-Weekly Rifapentine and Isoniazid in HIV-1-infected and HIV-1-uninfected Pregnant and Postpartum Women With Latent Tuberculosis Infection
Brief Title: Evaluating PK, Tolerability, and Safety of Rifapentine and Isoniazid in Pregnant and Postpartum Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT 2001; 12026 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2020-05

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — rifapentine; rifamycin SV; Isoniazid; Pyridoxine; Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (pregnant women enrolled in the second trimester) (Experimental): Participants received 12 directly observed once-weekly doses of RPT, INH, and pyridoxine (vitamin B6) at study entry and at 11 weekly follow-up visits.
  Interventions: Drug: Rifapentine (RPT); Drug: Isoniazid (INH); Dietary Supplement: Pyridoxine (vitamin B6)
- Cohort 2 (pregnant women enrolled in the third trimester) (Experimental): Participants received 12 directly observed once-weekly doses of RPT, INH, and pyridoxine (vitamin B6) at study entry and at 11 weekly follow-up visits.
  Interventions: Drug: Rifapentine (RPT); Drug: Isoniazid (INH); Dietary Supplement: Pyridoxine (vitamin B6)

INTERVENTIONS:
Drug: Rifapentine (RPT) — 900 mg of RPT
  Other Names: Rifamycin
Drug: Isoniazid (INH) — 900 mg of INH
  Other Names: isonicotinyl hydrazine,
Dietary Supplement: Pyridoxine (vitamin B6) — 25 mg to 100 mg of pyridoxine, based on the current local, national, or international dosing guidelines.
  Other Names: Vitamin B6

SUMMARY:
The purpose of this study was to evaluate the pharmacokinetics (PK), tolerability, and safety of once-weekly doses of rifapentine (RPT) and isoniazid (INH) in HIV-1-infected and HIV-1-uninfected pregnant and postpartum women with latent tuberculosis (TB).

DETAILED DESCRIPTION:
TB is a major cause of illness and death in women of reproductive age. Pregnant and postpartum women with latent TB are at higher risk of developing active TB. This study evaluated the pharmacokinetics, tolerability, and safety of 12 once-weekly doses of RPT and INH in HIV-1-infected and HIV-1-uninfected pregnant and postpartum women with latent TB.

This study enrolled HIV-1-infected and HIV-1-uninfected pregnant women with latent TB and their infants into two cohorts based on gestation. Cohort 1 participants were enrolled in their second trimester (greater than or equal to 14 to less than 28 weeks), and Cohort 2 participants were enrolled in their third trimester (greater than or equal to 28 to less than or equal to 34 weeks). All participants received 12 directly observed once-weekly doses of RPT, INH, and pyridoxine (vitamin B6) at study entry and at 11 weekly follow-up visits. Study researchers would perform an interim analysis to assess the PK of RPT during the study, and a dose adjustment could have been recommended based on this analysis.

Study visits occurred at days 0-3, once a week through week 11, and once a month until 24 weeks after delivery. Visits would include physical examinations, obstetrical exams, and blood collection. Infants were followed monthly until 24 weeks after birth.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years, or minimum age of consent according to locally applicable laws or regulations at screening, verified per site standard operating procedures (SOPs); and able and willing to provide written informed consent for study at screening
* At screening, evidence by ultrasound of a viable singleton pregnancy with an estimated gestational age at enrollment of greater than or equal to 14 weeks through less than or equal to 34 weeks as per screening ultrasound (see protocol for more information)
* Had at least one of the following risk factors for TB:

  * Per participant report, the participant was a household contact (see NOTE below) of a known active pulmonary TB patient
  * Per medical records, confirmation of HIV-1 infection (see protocol for more information) and a single positive tuberculin skin test (TST) or interferon gamma release assay (IGRA) at any time in the past. If not available in medical record, perform at screening.

NOTE: A household contact was defined as a person who currently lives or lived in the same dwelling unit and shares or shared the same housekeeping arrangements and who reported exposure within the past two years to an adult index case with pulmonary TB. Shared housekeeping arrangements were defined as sleeping under the same roof as the index TB case for at least seven consecutive days during the one month prior to the index case TB diagnosis.

* Documentation of HIV-1 infection status, or confirmation of HIV-1 infection status (if unknown or undocumented). Confirmation of HIV-1 infection was defined as positive results from two samples (described in the protocol) collected at different time points. All samples tested must be whole blood, serum, or plasma. As this study was being conducted under an IND, all test methods should be FDA-approved, if available. If FDA-approved methods were not available, test methods should be verified according to Good Clinical Laboratory Practice (GCLP) and approved by the IMPAACT Laboratory Center. More information on this criterion was available in the protocol.
* If HIV-1-infected, documented current prescription of efavirenz (EFV) + 2 nucleoside reverse transcriptase inhibitor (NRTI) regimen and reported taking regimen for at least two weeks prior to enrollment (regimens containing protease, integrase, or entry inhibitors were not permitted)
* Documented laboratory values obtained within 14 days prior to enrollment:

  * Hemoglobin greater than or equal to 7.5 g/dL
  * White blood cell count greater than or equal to 1500 cells/mm^3
  * Alanine transaminase (ALT) less than 2.5 times the upper limit of normal (ULN)
  * Total bilirubin less than 1.6 times the ULN
  * Absolute neutrophil count (ANC) greater than or equal to 750 cells/mm^3
  * Platelet count greater than or equal to 100,000/mm^3
* Per participant report at screening, intent to remain in the current geographical area of residence for the duration of the study
* Per participant report at screening, able to swallow whole tablets
* Per participant report, intention to keep the pregnancy
* Per participant report, willingness to permit infant to participate in the study

Exclusion Criteria:

* Evidence of confirmed or probable active TB disease per World Health Organization (WHO) symptom screen and confirmation by Gene Xpert, shielded chest x-ray, or sputum sample
* Participant report of personal history of INH- or rifampin-resistant, multi-drug resistant (MDR), or extensively drug-resistant (XDR) TB
* Participant report of personal history of active TB in the past 2 years
* Participant report of previous treatment for latent tuberculosis infection (LTBI)
* Household contact (as defined above) with known active MDR or XDR TB disease
* Known major fetal abnormality as detected on ultrasound
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation
* Known history of liver cirrhosis at any time prior to study entry
* Per participant report and/or medical records, evidence of acute clinical hepatitis, such as a combination of abdominal pain, jaundice, dark urine, and/or light stools within 90 days prior to entry
* Participant report and/or medical records of peripheral neuropathy Grade 2 or higher within 90 days prior to entry
* Current use or history of active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Participant report and/or clinical evidence of porphyria
* Any other condition that, in the opinion of the investigator of record (IoR)/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives, including taking the study medication
* Planned or current participation in an interventional drug study
* Current use of any prohibited or precautionary medications (see protocol for more information), including didanosine (DDI) or stavudine (D4T)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti S. Mathad, MD, MSc, Study Chair — Weill Medical College of Cornell University
Locations (5):
- Les Centres GHESKIO Clinical Research Site (GHESKIO-INLR) CRS, Port-au-Prince, Haiti
- Kenya Medical Research Institute / Walter Reed Project Clinical Research Center, Kericho CRS, Kericho, Kenya
- Malawi CRS, Lilongwe, Central Malawi, Malawi
- Siriraj Hospital ,Mahidol University NICHD CRS, Bangkok, Bangkoknoi, Thailand
- Harare Family Care CRS, Harare, Zimbabwe

REFERENCES:
- [Derived] Mathad JS, Savic R, Britto P, Jayachandran P, Wiesner L, Montepiedra G, Norman J, Zhang N, Townley E, Chakhtoura N, Bradford S, Patil S, Popson S, Chipato T, Rouzier V, Langat D, Chalermchockcharoentkit A, Kamthunzi P, Gupta A, Dooley KE. Pharmacokinetics and Safety of 3 Months of Weekly Rifapentine and Isoniazid for Tuberculosis Prevention in Pregnant Women. Clin Infect Dis. 2022 May 3;74(9):1604-1613. doi: 10.1093/cid/ciab665. PMID 34323955
- See also: Severity and laboratory tests will be graded per the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 2.0(dated November 2014 available on the RSC website) — http://rsc.tech-res.com/safetyandpharmacovigilance/
- See also: Requirements, definitions and methods for expedited reporting of adverse events (AEs) are outlined in Version 2.0 of the DAIDS EAE Manual — http://rsc.tech-res.com/safetyandpharmacovigilance/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on March 13, 2017 and accrual was completed on June 12, 2018 across the following sites: Siriraj Hospital, Mahidol University NIC (CRS 5115), Kenya Medical Research Institute/Walter Reed Project (CRS 5121), Malawi (CRS 12001), the Les Centres GHESKIO INLR (CRS 30022), and Harare Family Care (CRS 31890).
Period: Overall Study
Arm/Group | Cohort 1 (Pregnant Women Enrolled in the Second Trimester) | Cohort 2 (Pregnant Women Enrolled in the Third Trimester)
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Pregnant Women Enrolled in the Second Trimester) | Cohort 2 (Pregnant Women Enrolled in the Third Trimester) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 3 | 4
  Between 18 and 65 years | 24 | 22 | 46
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [22 to 33] | 27 [20 to 31] | 27 [20 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Non-Hispanic | 24 | 23 | 47
  Asian, Pacific Islander | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Haiti | 11 | 5 | 16
  Malawi | 2 | 1 | 3
  Zimbabwe | 9 | 12 | 21
  Kenya | 2 | 5 | 7
  Thailand | 1 | 2 | 3
HIV-1 status [Count of Participants; unit: Participants]
  HIV-1 uninfected | 15 | 15 | 30
  HIV-1 infected | 10 | 10 | 20
Absolute CD4 count [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: CD4 cell counts were assessed for HIV-1 infected mothers only
  cells/mm^3
    number analyzed (Participants) | 10 | 10 | 20
    (all) | 586 [415 to 846] | 489 [368 to 952] | 510 [390 to 877]
World Health Organization (WHO) clinical stage [Count of Participants; unit: Participants] — World Health Organization (WHO) produced WHO Disease Staging System for HIV Infection and Disease in Adults and Children. There are 4 stages of disease staging, 1 being the least severe and 4 being the most severe disease stage based on the HIV related symptoms and diagnoses. Please refer to the following web page for detailed staging criteria:
  https://www.who.int/hiv/pub/vct/hivstaging/en/ Population: WHO stages were assessed for HIV-1 infected mothers only
  Participants
    number analyzed (Participants) | 10 | 10 | 20
    Clinical Stage 1 | 10 | 10 | 20
    Clinical Stage 2 | 0 | 0 | 0
    Clinical Stage 3 | 0 | 0 | 0
    Clinical Stage 4 | 0 | 0 | 0
Weight [Median (Inter-Quartile Range); unit: kilograms] | 59 [55 to 66] | 61 [58 to 67] | 61 [56 to 67]
Gestational Age at Screening [Median (Inter-Quartile Range); unit: weeks] | 20 [16 to 24] | 30 [28 to 31] | 26 [20 to 30]
Mid-upper arm circumference (MUAC) [Median (Inter-Quartile Range); unit: centimeters] | 27 [25 to 31] | 27 [26 to 29] | 27 [25 to 30]
Serum glutamic-oxaloacetic transaminase (SGOT) [Median (Inter-Quartile Range); unit: units/L] | 21 [16 to 26] | 21 [18 to 23] | 21 [16 to 26]
Serum glutamic pyruvic transaminase (SGPT) [Median (Inter-Quartile Range); unit: units/L] | 17 [13 to 21] | 14 [11 to 17] | 15 [11 to 19]
Prothrombin Time result [Median (Inter-Quartile Range); unit: seconds] | 10 [10 to 11] | 11 [10 to 12] | 10 [10 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Clearance Relative to Bioavailability (CL/F) for Rifapentine (RPT) for Intensive and Sparse PK
Description: PK parameters were determined from plasma concentration-time profiles using a nonlinear mixed effects model (version 7.4; ICON PLC, Dublin, Ireland).
  * Developed a 1 compartment PK model with transit compartments for oral absorption
  * Calculated an average CL for all women in the 2nd trimester (cohort I) and all women in the 3rd trimester (cohort II)
Time Frame: Data used in the population PK analysis included the intensive PK visit (pre-dose (t0) and 0.5, 1, 2. 4, 5, 8, 12, 24, 48, 72 hours post-dose) and sparse PK visit (1, 4, 24, 48 hours post-dose).
Population: All participants with intensive and sparse PK results at all doses in all stages of pregnancy were used for analysis.
Measure: Mean (Inter-Quartile Range); unit: L/hr
Arm/Group | Cohort 1 (Pregnant Women Enrolled in the Second Trimester) | Cohort 2 (Pregnant Women Enrolled in the Third Trimester)
Number analyzed (Participants) | 24 | 25
L/hr | 1.4 [1.26 to 1.60] | 1.50 [1.25 to 1.66]

2. Primary Outcome: Clearance Relative to Bioavailability (CLmet/F) for Desacetyl Rifapentine (Des-RPT)
Description: PK parameters were determined from plasma concentration-time profiles using a nonlinear mixed effects model (version 7.4; ICON PLC, Dublin, Ireland).
  * Developed a 1 compartment PK model with transit compartments for oral absorption and a separate compartment for metabolite formation
  * Estimated a single des-RPT CLmet/F for the whole population Note: that the mean stated below is actually the value that is obtained from a population analysis and represents a population estimate with the relative standard error
Time Frame: as for outcome 1
Population: All participants with intensive and sparse PK results at all doses in all stages of pregnancy were used for analysis.
Measure: Mean (Standard Error); unit: L/hr
Groups:
- All Cohorts: Combined for all women in Second and Third Trimester of pregnancy
Arm/Group | All Cohorts
Number analyzed (Participants) | 49
L/hr | 2.82 (7)

3. Primary Outcome: Absorption Rate Constant (ka) for Rifapentine (RPT)
Description: PK parameters were determined from plasma concentration-time profiles using a nonlinear mixed effects model (version 7.4; ICON PLC, Dublin, Ireland).
  * Developed a 1 compartment PK model with transit compartments for oral absorption
  * Estimated the transit compartment rate constant (ktr), which is synonymous with the absorption constant (ka), for the whole population Note that the mean stated below is actually the value that is obtained from a population analysis and represents a population estimate
Time Frame: as for outcome 1
Population: All participants with intensive and sparse PK results at all doses in all stages of pregnancy were used for analysis.
Measure: Mean (Standard Error); unit: hr-1
Arm/Group | All Cohorts
Number analyzed (Participants) | 49
hr-1 | 1.43 (NA) — The absorption rate is calculated from another estimated parameter and hence there is no Relative Standard Error to report and hence the value of N/A was entered.

4. Primary Outcome: Volume of Distribution Relative to Bioavailability (Vc/F) for Rifapentine (RPT)
Description: PK parameters were determined from plasma concentration-time profiles using a nonlinear mixed effects model (version 7.4; ICON PLC, Dublin, Ireland).
  * Developed a 1 compartment PK model with transit compartments for oral absorption
  * Estimated a single RPT Vc/F for for the whole population Note: that the mean stated below is actually the value that is obtained from a population analysis and represents a population estimate with the relative standard error
Time Frame: as for outcome 1
Population: All participants with intensive and sparse PK results at all doses in all stages of pregnancy were used for analysis.
Measure: Mean (Standard Error); unit: L
Arm/Group | All Cohorts
Number analyzed (Participants) | 49
L | 30.1 (5)

5. Primary Outcome: Incidence of Related Serious Adverse Events (SAEs) in Pregnant and Postpartum Women Taking Once-weekly RPT + INH
Description: At entry and follow-up, all lab results, sign and symptoms, and diagnoses were recorded. Also, during follow-up grade 2 events related to pregnancy complications, hepatotoxicity, hemorrhage, or peripheral neuropathy, and all grade 3 or events that resulted in discontinuation of study drug regimen, and that met criteria for EAE reporting would further be evaluated and recorded. The DAIDS Table for Grading Adult and Pediatric Adverse Events (V 2.0) and Expedited AE Manual (V 2.0) were used.
Time Frame: Measured from entry through participants' last study visit at 24 weeks after delivery
Population: All participants enrolled in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Pregnant Women Enrolled in the Second Trimester) | Cohort 2 (Pregnant Women Enrolled in the Third Trimester)
Number analyzed (Participants) | 25 | 25
Participants | 0 | 0

6. Primary Outcome: Percentage of Participants With Grade 2 Adverse Events (AEs) Judged to be Related to Study Drug Regimen
Description: At entry and follow-up, all lab results, sign and symptoms, and diagnoses were recorded. Also, during follow-up grade 2 events related to pregnancy complications, hepatotoxicity, hemorrhage, or peripheral neuropathy, and all grade 3 or events that resulted in discontinuation of study drug regimen, and that met criteria for EAE reporting would further be evaluated and recorded. The DAIDS Table for Grading Adult and Pediatric Adverse Events (V 2.0) and Expedited AE Manual (V 2.0) and were used.
Time Frame: Measured from study entry through participants' last study visit at 24 weeks after delivery
Population: All participant enrolled on the study
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Cohort 1 (Pregnant Women Enrolled in the Second Trimester) | Cohort 2 (Pregnant Women Enrolled in the Third Trimester)
Number analyzed (Participants) | 25 | 25
percent of participants | 4 [0.1 to 20] | 0 [0 to 14]

7. Primary Outcome: Percentage of Participants With All Grade 3 and 4 AEs
Description: as for outcome 5
Time Frame: Measured from study entry through participants' last study visit at 24 weeks after delivery
Population: All participants enrolled on the study
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Cohort 1 (Pregnant Women Enrolled in the Second Trimester) | Cohort 2 (Pregnant Women Enrolled in the Third Trimester)
Number analyzed (Participants) | 25 | 25
percent of participants | 20 [7 to 41] | 16 [5 to 36]

8. Primary Outcome: Percentage of Participants With All Serious AEs
Description: as for outcome 5
Time Frame: Measured from study entry through participants' last study visit at 24 weeks after delivery
Population: All participants enrolled on the study
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Cohort 1 (Pregnant Women Enrolled in the Second Trimester) | Cohort 2 (Pregnant Women Enrolled in the Third Trimester)
Number analyzed (Participants) | 25 | 25
percent of participants | 8 [1 to 26] | 12 [3 to 31]

9. Primary Outcome: Percentage of Participants With All AEs Leading to Permanent Discontinuation of Study Drug Regimen (i.e., RPT, INH, and Pyridoxine)
Description: as for outcome 5
Time Frame: Measured from study entry through participants' last study treatment dispensation (approximately for 12 weeks)
Population: All participants enrolled on the study
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Cohort 1 (Pregnant Women Enrolled in the Second Trimester) | Cohort 2 (Pregnant Women Enrolled in the Third Trimester)
Number analyzed (Participants) | 25 | 25
percent of participants | 0 [0 to 14] | 0 [0 to 14]

10. Primary Outcome: Percentage of Participants With Related Serious Adverse Events (AEs) in Infants Born to Women Taking Once-weekly RPT + INH
Description: as for outcome 5
Time Frame: Measured from birth through infants' last study visit at 24 weeks after birth
Population: For the 49 live born infants to the women enrolled on the study
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- Cohort 1 (Infants Born to Women Enrolled in Second Trimester); Cohort 2 (Infants Born to Women Enrolled in Third Trimester): Infants born to women who received 12 directly observed once-weekly doses of RPT, INH, and pyridoxine (vitamin B6) at study entry and at 11 weekly follow-up visits.
Arm/Group | Cohort 1 (Infants Born to Women Enrolled in Second Trimester) | Cohort 2 (Infants Born to Women Enrolled in Third Trimester)
Number analyzed (Participants) | 24 | 25
percent of participants | 0 [0 to 14] | 0 [0 to 14]

11. Secondary Outcome: Clearance Relative to Bioavailability (CL/F) for Rifapentine (RPT)
Description: PK parameters from postpartum women were determined from plasma concentration-time profiles using a nonlinear mixed effects model (version 7.4; ICON PLC, Dublin, Ireland).
  * Developed a 1 compartment PK model with transit compartments for oral absorption
  * Calculated an average CL for all post-partum individuals
Time Frame: Data used in the population PK analysis for postpartum women included the intensive PK visit (pre-dose (t0) and 0.5, 1, 2. 4, 5, 8, 12, 24, 48, 72 hours post-dose) and sparse PK visit (1, 4, 24, 48 hours post-dose).
Population: All participants with intensive and sparse PK results at all doses postpartum were used for analysis.
Measure: Mean (Inter-Quartile Range); unit: L/hr
Groups:
- All Cohorts: All postpartum women
Arm/Group | All Cohorts
Number analyzed (Participants) | 22
L/hr | 1.64 [1.6 to 1.68]

12. Secondary Outcome: Area Under the Curve From 0 to 24 Hours (AUC0-24) for RPT and Area Under the Curve From 0 to 24 Hours (AUC0-24) for Des-RPT Pregnant Women in 2nd and 3rd Trimester
Description: PK parameters were determined from plasma concentration-time profiles using a nonlinear mixed effects model (version 7.4; ICON PLC, Dublin, Ireland).
  * Developed a 1 compartment PK model with transit compartments for oral absorption
  * Obtained AUC by model-based integration
Time Frame: as for outcome 1
Population: All participants with intensive and sparse PK results for RPT at all doses in all stages of pregnancy were used for analysis
Measure: Mean (Inter-Quartile Range); unit: hour*mg/L
Arm/Group | Cohort 1 (Pregnant Women Enrolled in the Second Trimester) | Cohort 2 (Pregnant Women Enrolled in the Third Trimester)
Number analyzed (Participants) | 22 | 19
hour*mg/L
  AUC (0-24) for RPT | 424.7 [341.7 to 514.1] | 406.8 [334.8 to 471.7]
  AUC (0-24) for des-RPT | 158.7 [118.9 to 184.3] | 153.7 [123.1 to 186.4]

13. Secondary Outcome: Maximum Concentration (Cmax) for RPT Maximum Concentration (Cmax) for Des-RPT Pregnant Women in 2nd and 3rd Trimester
Description: PK parameters were determined from plasma concentration-time profiles using a nonlinear mixed effects model (version 7.4; ICON PLC, Dublin, Ireland).
  * Developed a 1 compartment PK model with transit compartments for oral absorption
  * Obtained Cmax by model-based estimation
Time Frame: as for outcome 1
Population: as for outcome 12
Measure: Mean (Inter-Quartile Range); unit: mg/L
Arm/Group | Cohort 1 (Pregnant Women Enrolled in the Second Trimester) | Cohort 2 (Pregnant Women Enrolled in the Third Trimester)
Number analyzed (Participants) | 22 | 19
mg/L
  Cmax for RPT | 30.2 [25.1 to 36.1] | 28.6 [24.7 to 32.1]
  Cmax for des-RPT | 8.76 [5.91 to 10.8] | 8.50 [6.82 to 10.0]

14. Secondary Outcome: Maximum Concentration (Cmin) for RPT and Maximum Concentration (Cmin) for Des-RPT Pregnant Women in 2nd and 3rd Trimester
Description: PK parameters were determined from plasma concentration-time profiles using a nonlinear mixed effects model (version 7.4; ICON PLC, Dublin, Ireland).
  * Developed a 1 compartment PK model with transit compartments for oral absorption
  * Obtained Cmin by model-based estimation
Time Frame: as for outcome 1
Population: as for outcome 12
Measure: Mean (Inter-Quartile Range); unit: mg/L
Arm/Group | Cohort 1 (Pregnant Women Enrolled in the Second Trimester) | Cohort 2 (Pregnant Women Enrolled in the Third Trimester)
Number analyzed (Participants) | 23 | 25
mg/L
  Cmin for RPT | 1.45 [0.84 to 1.98] | 1.58 [0.66 to 2.29]
  Cmin for des-RPT | 1.06 [0.63 to 1.25] | 1.20 [0.79 to 1.74]

15. Secondary Outcome: Cord Blood Concentrations of Rifapentine (RPT) Among Infants
Description: Cord blood concentrations were summarized using using R (version 3.5.1).
Time Frame: at delivery - (within 3 days of life for infants)
Population: All infants with available concentration data born to women on the study
Measure: Mean (Inter-Quartile Range); unit: mcg/mL
Groups:
- All Cohorts: Combined for all infants born to women in Second and Third Trimester of pregnancy
Arm/Group | All Cohorts
Number analyzed (Participants) | 5
mcg/mL | 2.97 [1.94 to 4.26]

16. Secondary Outcome: Plasma Concentrations of Rifapentine (RPT) Among Infants
Description: Plasma concentrations were summarized using using R (version 3.5.1).
Time Frame: at delivery - (within 3 days of life for infants).
Population: All infants with available concentrations born to women on the study
Measure: Mean (Inter-Quartile Range); unit: mcg/mL
Arm/Group | All Cohorts
Number analyzed (Participants) | 8
mcg/mL | 2.47 [1.49 to 3.30]

17. Secondary Outcome: Cord Blood Concentrations of Desacetyl Rifapentine (Des-RPT) Among Infants
Description: Cord blood concentrations were summarized using using R (version 3.5.1).
Time Frame: at delivery (within 3 days of life for infants).
Population: All infants with available concentrations born to women on the study
Measure: Mean (Inter-Quartile Range); unit: mcg/mL
Arm/Group | All Cohorts
Number analyzed (Participants) | 5
mcg/mL | 3.24 [1.03 to 5.17]

18. Secondary Outcome: Plasma Concentrations of Desacetyl Rifapentine (Des-RPT) Among Infants
Description: Plasma blood concentrations were summarized using using R (version 3.5.1).
Time Frame: at delivery - (within 3 days of life for infants).
Population: All infants with available concentrations born to women on the study
Measure: Mean (Inter-Quartile Range); unit: mcg/mL
Arm/Group | All Cohorts
Number analyzed (Participants) | 8
mcg/mL | 5.31 [3.73 to 7.37]

19. Secondary Outcome: Number of Participants With Discontinuation of Study Drug Due to Intolerance (Tolerability of Study Drug Regimen - i.e., RPT, INH, and Pyridoxine)
Description: At entry and follow-up, all lab results, sign and symptoms, and diagnoses will be recorded. Also, during follow-up grade 2 events related to pregnancy complications, hepatotoxicity, hemorrhage, or peripheral neuropathy, and all grade 3 or events that result in discontinuation of study drug regimen, and that meet criteria for EAE reporting will be further evaluated and recorded. The DAIDS Table for Grading Adult and Pediatric Adverse Events (V 2.0) and Expedited AE Manual (V 2.0) were used.
Time Frame: Measured from study entry through participants' last study visit at 24 weeks after delivery
Population: All participants enrolled on the study
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Pregnant Women Enrolled in the Second Trimester) | Cohort 2 (Pregnant Women Enrolled in the Third Trimester)
Number analyzed (Participants) | 25 | 25
Participants | 0 | 0

20. Secondary Outcome: Number of Mothers With Active TB up to 24 Weeks Postpartum
Description: Based on site-specified confirmatory TB test. If women and infants were diagnosed with active TB during study they would be referred to local care for TB management and treatment.
Time Frame: Measured from study entry through participants' last study visit at 24 weeks after delivery
Population: All participants enrolled on the study
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Pregnant Women Enrolled in the Second Trimester) | Cohort 2 (Pregnant Women Enrolled in the Third Trimester)
Number analyzed (Participants) | 25 | 25
Participants | 0 | 0

21. Secondary Outcome: Number of Infants With Active TB up to 24 Weeks of Life
Description: as for outcome 20
Time Frame: Measured from birth through participants' last study visit at 24 weeks after delivery
Population: All live born infants enrolled on the study
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1(Infants Born to Women Enrolled in Second Trimester): Participants received 12 directly observed once-weekly doses of RPT, INH, and pyridoxine (vitamin B6) at study entry and at 11 weekly follow-up visits.
- Cohort 2 (Infants Born to Women Enrolled in Third Trimester): Participants will receive 12 directly observed once-weekly doses of RPT, INH, and pyridoxine (vitamin B6) at study entry and at 11 weekly follow-up visits.
Arm/Group | Cohort 1(Infants Born to Women Enrolled in Second Trimester) | Cohort 2 (Infants Born to Women Enrolled in Third Trimester)
Number analyzed (Participants) | 24 | 25
Participants | 0 | 0

22. Secondary Outcome: Clearance (CL/F) of INH
Description: PK parameters were determined from plasma concentration-time profiles using a nonlinear mixed effects model (version 7.4; ICON PLC, Dublin, Ireland).
  * Developed a 1 compartment PK model with 2 mixtures to characterize subpopulations based on acetylation status
  * Estimated a separate INH CL/F based on acetylation status (fast, slow)
Time Frame: as for outcome 1
Population: All participants with intensive and sparse PK results at all doses in all stages of pregnancy were used for analysis Note: the mean reported below is actually the value obtained from a population analysis and represents a population estimate with relative standard error
Measure: Mean (Standard Error); unit: L/hr
Groups:
- All Cohorts: All participants with intensive and sparse PK results at all doses in all stages of pregnancy were used for analysis
Arm/Group | All Cohorts
Number analyzed (Participants) | 49
L/hr
  CL/F (slow acetylators) | 8.98 (47)
  CL/F (fast acetylators) | 32.7 (10)

23. Secondary Outcome: Absorption (ka) of INH
Description: PK parameters were determined from plasma concentration-time profiles using a nonlinear mixed effects model (version 7.4; ICON PLC, Dublin, Ireland).
  • Estimated a single absorption rate constant (ka) for the whole population
Time Frame: as for outcome 1
Population: as for outcome 22
Measure: Mean (Standard Error); unit: hr-1
Arm/Group | All Cohorts
Number analyzed (Participants) | 49
hr-1 | 1.74 (49)

24. Secondary Outcome: Volume of Distribution of INH
Description: PK parameters were determined from plasma concentration-time profiles using a nonlinear mixed effects model (version 7.4; ICON PLC, Dublin, Ireland).
  • Estimated a single INH Vc/F for the whole population
Time Frame: as for outcome 1
Population: as for outcome 22
Measure: Mean (Standard Error); unit: L
Arm/Group | All Cohorts
Number analyzed (Participants) | 49
L | 107 (12)

ADVERSE EVENTS:
Time Frame: Measured from study entry through participants last study visit at 24 weeks after delivery
Description: At entry and follow-up, all lab results, sign and symptoms, and diagnoses were recorded. Also, during follow-up grade 2 events related to pregnancy complications, hepatotoxicity, hemorrhage, or peripheral neuropathy, and all grade 3 or events that resulted in discontinuation of study drug regimen, and that met criteria for EAE reporting would further be evaluated and recorded. The DAIDS Table for Grading Adult and Pediatric Adverse Events (V 2.0) and Expedited AE Manual (V 2.0) were used.
Groups:
- Cohort 1 (Pregnant Women Enrolled in Their Second Trimester); Cohort 2 (Pregnant Women Enrolled in Their Third Trimester): Participants received 12 directly observed once-weekly doses of RPT, INH, and pyridoxine (vitamin B6) at study entry and at 11 weekly follow-up visits.
Arm/Group | Cohort 1 (Pregnant Women Enrolled in Their Second Trimester) | Cohort 2 (Pregnant Women Enrolled in Their Third Trimester)
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25 | 3/25
Other Adverse Events (participants affected / at risk) | 24/25 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Pregnant Women Enrolled in Their Second Trimester) (N=25) | Cohort 2 (Pregnant Women Enrolled in Their Third Trimester) (N=25)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Pregnant Women Enrolled in Their Second Trimester) (N=25) | Cohort 2 (Pregnant Women Enrolled in Their Third Trimester) (N=25)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 | 0
Palpitations (Cardiac disorders) | 2 | 0
Eye pain (Eye disorders) | 2 | 1
Ocular hyperaemia (Eye disorders) | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Abdominal pain lower (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 5 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Chest pain (General disorders) | 2 | 1
Malaise (General disorders) | 5 | 0
Oedema peripheral (General disorders) | 3 | 1
Pyrexia (General disorders) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 2
Vulvovaginal candidiasis (Infections and infestations) | 2 | 3
Incision site pain (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 4 | 5
Aspartate aminotransferase increased (Investigations) | 6 | 7
Blood albumin decreased (Investigations) | 20 | 21
Blood bilirubin increased (Investigations) | 2 | 0
Blood pressure increased (Investigations) | 5 | 3
Haemoglobin decreased (Investigations) | 15 | 10
Platelet count decreased (Investigations) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Headache (Nervous system disorders) | 6 | 5
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Dysuria (Renal and urinary disorders) | 4 | 1
Pelvic pain (Reproductive system and breast disorders) | 8 | 4
Vaginal discharge (Reproductive system and breast disorders) | 2 | 4
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (3):
  • Study Protocol (2015-11-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT02651259/Prot_002.pdf
  • Statistical Analysis Plan: Final Safety Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT02651259/SAP_000.pdf
  • Statistical Analysis Plan: Final PK Statistical Analysis Plan (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT02651259/SAP_001.pdf